CLINICAL TRIAL: NCT02766062
Title: Effects of Propofol and Sevoflurane on Early Postoperative Cognitive Dysfunction in Elderly Patients With Metabolic Syndrome
Brief Title: Effects of Propofol and Sevoflurane on Early POCD in Elderly Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NZ1651
Record Dates: First submitted 2016-05-01; First posted 2016-05-09 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Complications
Keywords: Postoperative cognitive dysfunction; metabolic syndrome; propofol; sevoflurane
MeSH Terms: conditions — Postoperative Complications; Postoperative Cognitive Complications; Metabolic Syndrome | interventions — ANAPC16 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol group (Active Comparator): Patients with metabolic syndrome were randomly assigned to receive propofol anesthesia
  Interventions: Other: metabolic syndrome
- sevoflurane group (Active Comparator): Patients with metabolic syndrome were randomly assigned to receive sevoflurane anesthesia
  Interventions: Other: metabolic syndrome

INTERVENTIONS:
Other: metabolic syndrome — metabolic syndrome

SUMMARY:
The purpose of this study is to investigate propofol versus sevoflurane anesthesia on the effects of early postoperative cognitive function in elderly patients with metabolic syndrome.

DETAILED DESCRIPTION:
By now, a series risk factors of cardiovascular diseases, which are also related to the development of postoperative cognitive dysfunction (POCD), are becoming more common.The investigators don't know whether propofol based anesthesia has a more severe impact on early postoperative cognitive function than sevoflurane in elderly patients with metabolic syndrome. In this study, the investigators want to investigate propofol versus sevoflurane anesthesia on the effects of early postoperative cognitive function in elderly patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥60 years;
* ASAⅡor Ⅲ
* noncardiac surgery and nonneural surgery

Exclusion Criteria:

* Mini Mental State Examination [MMSE] score too low
* chronic alcoho and drug abuse
* disturbed renal and liver function
* history of a cerebrovascular accident
* permanent ventricular pacing
* preoperative cognitive deficits
* lack of cooperation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with Postoperative cognitive dysfunction (POCD) as assessed by Mini-Mental State Examination (MMSE) score in propofol group and sevoflurane group | up to 7days postoperatively

IPD SHARING:
Plan to Share IPD: No
safety